CLINICAL TRIAL: NCT04236986
Title: Imaging the Neuroimmune System in PTSD With PET
Brief Title: Imaging the Neuroimmune System in PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelly Cosgrove, Associate Professor, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000020347; 1R01MH110674-01A1 (NIH)
Record Dates: First submitted 2020-01-11; First posted 2020-01-22 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Neuroimmune System; Lipopolysaccharide
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: All subjects will complete a baseline PET [11C]PBR28 scan. A subset of subjects will complete a second PET [11C]PBR28 scan 3-hours after systemic LPS challenge (1.0 ng/kg; IV).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baseline [11C]PBR28 PET Scan (No Intervention): Subjects will complete a 120-minute baseline [11C]PBR28 PET scan.
- Post-LPS [11C]PBR28 PET Scan (Experimental): Subjects will complete a second120-minute [11C]PBR28 PET scan 3-hours after LPS administration (1.0ng/kg; IV)
  Interventions: Drug: Lipopolysaccharide

INTERVENTIONS:
Drug: Lipopolysaccharide — LPS will be administered intravenously (1.0ng/kg; IV)
  Other Names: LPS
  Arms: Post-LPS [11C]PBR28 PET Scan

SUMMARY:
In this study, individuals with and without post-traumatic stress disorder (PTSD) will undergo one positron emission tomography (PET) scan using the radiotracer [11C]PBR28, which binds to the 18kDa translocator protein (TSPO). A subset of individuals who complete the first PET [11C]PBR28 scan will be invited to complete an inflammatory challenge and second PET [11C]PBR28 scan. Approximately 3 hours prior to the second [11C]PBR28 PET scan, lipopolysaccharide (LPS; endotoxin) will be administered to evoke a robust neuroimmune response. Subjects will also undergo behavioral and cognitive testing. Vital signs, subjective response, and peripheral biomarker levels will be assayed periodically throughout the experimental session.

Specific aims: 1) Determine if individuals with PTSD exhibit neuroimmune system disruption relative to well-matched comparators at baseline. 2) Determine if individuals with PTSD exhibit a disrupted neuroimmune response after a classical immune stimulus relative to well-matched comparators. 3) Determine if LPS differentially alters cognitive function, subjective response, or physiological markers in individuals with PTSD compared to well-matched comparators.

Hypothesis: Individuals with PTSD will exhibit a suppressed neuroimmune system at baseline and an attenuated neuroimmune response following LPS challenge, relative to matched trauma controls.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18-55 years
2. Subjects with PTSD will have a primary, current diagnosis of PTSD according to DSM-V criteria (i.e., CAPS-5 ascertained diagnosis)
3. Able to read and write English and to provide voluntary, written informed consent

Exclusion Criteria:

1. Current medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology including COPD, anemia, uncontrolled daily asthma or asthma requiring the use of an inhaler more than 1x/week with an ACT score below 20. [We will not exclude individuals taking SSRIs and TRIs due to high prevalence of use within the PTSD population and due to evidence suggesting no effect of these drug classes on endotoxin response].
2. Past or current neurological disorder or disorders affecting the brain including but not limited to multiple sclerosis, history of stroke, brain tumors, traumatic brain injury with loss of consciousness, seizure disorder
3. Current or regular use of over-the-counter medication that may affect the immune system
4. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD
5. Contraindications to MRI such as claustrophobia or metal in their body
6. Individuals who are classified as "low binders" for the rs6971 polymorphism (<10% of the population)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347: We will recruit men and women aged 18-55 who have been exposed to trauma without PTSD into the study. Men and women, aged 18-55 years, any race, with a history of trauma exposure.
  Trauma-exposed controls will have a CAPS-5 score of 0-22 (no/minimal to mild/subthreshold symptoms) Able to read and write English and to provide voluntary, written informed consent
- PTSD Controls for HIC 2000020347: We will recruit men and women aged 18-55 who have been exposed to trauma with PTSD into the study. Men and women, aged 18-55 years, any race, with a history of PTSD, Subjects with posttraumatic stress disorder (PTSD) will have a primary, current diagnosis of PTSD according to DSM-V criteria (i.e., CAPS-5 ascertained diagnosis) Able to read and write English and to provide voluntary, written informed consent
Period: Overall Study
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Started | 18 | 16
Completed | 15 | 15
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347 | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 subjects withdrew from HC population and 1 subject from PTSD population withdrew, prior to second PET scan and LPS injection.
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    Female | 4 | 6 | 10
    Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 healthy controls and 1 PTSD participant declined to continue/withdrew from study prior to second PET scan/LPS
  Participants
    number analyzed (Participants) | 15 | 15 | 30
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 5 | 8
    White | 7 | 7 | 14
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Baseline TSPO Availability
Description: Time-activity curves will be extracted from brain regions of interest and analyzed using multilinear analysis-1 (t*=30) incorporating the metabolite-corrected arterial input function to yield [11C]PBR28 total volumes of distribution (VT) across brain regions.
Time Frame: Before LPS administration (baseline)
Measure: Mean (Standard Deviation); unit: mL/cm3
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 15 | 15
mL/cm3
  Amygdala | 5.11 (.85) | 4.75 (1.35)
  insula | 5.07 (.85) | 4.38 (1.1)
  vmPFC | 5.33 (.9) | 5.33 (1.16)
  hippocampus | 4.89 (.78) | 4.38 (1.1)

2. Primary Outcome: Post-LPS TSPO Availability
Description: as for outcome 1
Time Frame: 3-hours after LPS administration (1.0 ng/kg; IV)
Measure: Mean (Standard Deviation); unit: mL/cm3
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 15 | 15
mL/cm3
  Amygdala | 7.2 (1.37) | 6.07 (2.12)
  Hippocampus | 6.82 (.87) | 5.66 (1.8)
  Insula | 7.14 (1.3) | 7.14 (2.1)
  vmPFC | 7.73 (1.6) | 7.73 (1.8)

3. Secondary Outcome: Baseline Visual Attention
Description: Visual attention: response latency to identify card color (log10(ms); higher ~ worse attention).
Time Frame: Before LPS administration
Measure: Mean (Full Range); unit: log10(ms)
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
log10(ms) | 2.624842444 [2.457448 to 2.951719] | 6.877150091 [2.312753 to 50]

4. Secondary Outcome: Post-LPS Visual Attention
Description: Visual attention: response latency to identify card color (log10(ms); higher ~ worse attention).
Time Frame: Approximately ~1-hour after LPS administration
Measure: Mean (Full Range); unit: log10(ms)
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
log10(ms) | 2.54493925 [2.3893 to 2.713619] | 2.6069589 [2.333067 to 2.764084]

5. Secondary Outcome: Baseline Visual Learning
Description: Visual learning: % of correctly identified repeat cards (arcsine(% correct); higher values ~ better learning).
Time Frame: Before LPS administration
Measure: Mean (Full Range); unit: percentage of correct responses
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
percentage of correct responses | 0.926197556 [0 to 1.306618] | 1.005693 [0.63029 to 1.336154]

6. Secondary Outcome: Post-LPS Visual Learning
Description: Visual learning: % of correctly identified repeat cards (arcsine(% correct); higher values ~ better learning).
Time Frame: Approximately ~1-hour after LPS administration
Measure: Mean (Full Range); unit: percentage of correct responses
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
percentage of correct responses | 0.98078875 [0.82031 to 1.115727] | 0.9055107 [0.61548 to 1.209429]

7. Secondary Outcome: Baseline Verbal Memory
Description: Verbal memory: summed number of correctly recalled items from a grocery list (over 3 trials). Each trial is not calculated individually. The reported value is the sum of all three trials.
Time Frame: Before LPS administration
Measure: Mean (Full Range); unit: Number of correct responses
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
Number of correct responses | 29.11111111 [22 to 35] | 27.45454545 [9 to 41]

8. Secondary Outcome: Post-LPS Verbal Memory
Description: Verbal memory: summed # of correctly recalled items from a grocery list (over 3 trials). Each trial is not calculated individually. The reported value is the sum of all three trials.
Time Frame: Approximately ~1-hour after LPS administration
Measure: Mean (Full Range); unit: Number of correct responses
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
Number of correct responses | 26.75 [18 to 31] | 25.7 [18 to 33]

9. Secondary Outcome: Baseline Executive Function
Description: Executive function: summed number of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function).
Time Frame: Before LPS administration
Measure: Mean (Full Range); unit: Number of errors
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
Number of errors | 51.11111111 [28 to 74] | 45.36363636 [0 to 103]

10. Secondary Outcome: Post-LPS Executive Function
Description: Executive function: summed number of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function).
Time Frame: Approximately ~1-hour after LPS administration
Measure: Mean (Full Range); unit: Number of errors
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
Number of errors | 57.5 [25 to 99] | 60.4 [34 to 111]

11. Secondary Outcome: Baseline Visual-Motor Processing Speed
Description: Visual-motor processing speed: response latency to detect a card flipped over (log10(ms); higher ~ worse processing speed).
Time Frame: Before LPS administration
Measure: Mean (Full Range); unit: log10(ms)
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
log10(ms) | 2.415812111 [0 to 2.878009] | 5.285026273 [2.54562 to 31]

12. Secondary Outcome: Post-LPS Visual-Motor Processing Speed
Description: as for outcome 11
Time Frame: Approximately ~1-hour after LPS administration
Measure: Mean (Full Range); unit: log10(ms)
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 9 | 13
log10(ms) | 2.74042025 [2.562187 to 2.859766] | 2.7598859 [2.54562 to 2.97832]

13. Secondary Outcome: Baseline Social Cognition
Description: Social cognition: response latency to identify the mismatched facial expression based on its emotional content (ms; log10; higher ~ worse social cognition).
Time Frame: Before LPS administration
Population: Data were not collected.
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Post-LPS Social Cognition
Description: as for outcome 13
Time Frame: Approximately ~1-hour after LPS administration
Population: Data were not collected.
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will be followed for 1 month after LPS injection and second PET scan.
Description: this study will be monitored every 6 months by a Data Safety Monitoring Board (DSMB). Adequate surveillance and protections will be put in place to discover adverse events promptly and keep their effects to a minimum. There is an established DSMB at the Yale PET Center that meets every 6 months.
  Expected and Unexpected Adverse Events will be recorded according to PET Center and NIH guidelines
Arm/Group | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 | PTSD Controls for HIC 2000020347
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 1/18 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls AKA Trauma Exposed Individuals Without PTSD For HIC 2000020347 (N=18) | PTSD Controls for HIC 2000020347 (N=16)
Dull ache Loose Bowels (General disorders) | 1 (1) | 0 (0) — Dull ache and loose bowels(diarrhea) post aline placement 2022-01-28, Date confirmed 02-02-2022 Self Resolved. Ache most likely attributed to aline placement. Loose bowels self resolved, cause unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT04236986/Prot_SAP_000.pdf
  • Informed Consent Form: ICF form 4 (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04236986/ICF_001.pdf
  • Informed Consent Form: ICF form 1 2 5 (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04236986/ICF_002.pdf